CLINICAL TRIAL: NCT03448471
Title: Pulmonary and Extra-pulmonary Characteristics in Severe-fatigued Allogeneic Hematopoietic Stem Cell Transplantation Recipients
Brief Title: Severe Fatigue in Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof., Gazi University
Other Study IDs: GaziUniversity4
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Stem Cell Transplantation; Fatigue
Keywords: stem cell transplantation; Fatigue; muscle strength; exercise capacity; Depression; Quality of Life
MeSH Terms: conditions — Fatigue; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: severe-fatigued recipients: These recipients had Fatigue Severity Scale score ≥36. All recipients evaluated with similar methods. Meaurements were Pulmonary function tests, Respiratory muscle strength, Peripheral muscle strength, Functional exercise capacity, Dyspnea, Fatigue, Depression and Quality of life.
- Group 2: non-severe-fatigued recipients: These recipients had Fatigue Severity Scale score <36. All recipients evaluated with similar methods. Meaurements were Pulmonary function tests, Respiratory muscle strength, Peripheral muscle strength, Functional exercise capacity, Dyspnea, Fatigue, Depression and Quality of life.

SUMMARY:
Fatigue is a common symptom during allogeneic-hematopoietic stem cell transplantation (allo-HSCT). However, effects of severe fatigue on pulmonary functions, blood cells, dyspnea, muscle strength, exercise capacity, depression and quality of life (QOL) in allo-HSCT recipients are still unknown.

DETAILED DESCRIPTION:
Fatigue is the most complained side effect that may last for months or even years after treatment ends in patients with cancer. Cancer-related fatigue is described as 'a distressing, persistent, subjective sense of physical, emotional and/or cognitive tiredness or exhaustion related to cancer or cancer treatment that is not proportional to recent activity and interferes with usual functioning'. The cancer-related fatigue observed in 80% of cancer patients received chemotherapy and/or radiotherapy, yet underlying mechanism of cancer-related fatigue is not still clearly explained.

Hematological malignancy itself and its treatments including chemotherapy, radiotherapy, surgery, medical treatment and/or allogeneic or autologous hematopoietic stem cell transplantation cause lots of early and late adverse effects such as appetite loss, nausea and vomiting, diarrhea, fatigue, sleep disturbance, pain, cardiopulmonary and neuromuscular deconditioning, impairments in mobility, muscle weakness and increased risk of fall.

Hematopoietic stem cells collected from bone marrow, peripheral blood or umbilical cord blood of healthy donors are infused into allogeneic hematopoietic stem cell transplantation (allogeneic-HSCT) recipients with hematological malignancy. Allogeneic-HSCT is highly associated with transplant-related mortality, morbidity, graft-versus host disease and another various complications. Because of the above-mentioned risks, recipients and their caregivers are required to remain close to transplant center in the acute phase of transplantation, approximately 100 days. As a consequence, hematopoietic stem cell transplantation has a negative impact on quality of life in recipients and their caregivers who report fatigue, sleep and sexual problems and emotional distress. Especially fatigue is a destructive symptom for recipients, exists before hematopoietic stem cell transplantation and further deteriorates during the first three weeks after hematopoietic stem cell transplantation. Moreover baseline fatigue severity continues until one year after hematopoietic stem cell transplantation.

Although fatigue has been one of the most intensely experienced symptoms by allogeneic-HSCT recipients, no study has compared pulmonary functions, albumin-hemoglobin-white blood cell levels, dyspnea, respiratory and peripheral muscle strength, submaximal exercise capacity, depression and quality of life between severe-fatigued and non-severe-fatigued allogeneic-HSCT recipients, yet. Therefore investigators aimed to compare the effects of severe fatigue on aforementioned outcomes in recipients.

ELIGIBILITY:
Inclusion Criteria:

* being an hematopoietic stem cell transplantation recipient during the intermediate/late post-transplant phase (>100 days),
* 18-65 years of age
* under standard medications.

Exclusion Criteria:

* having a cognitive disorder,
* orthopedic or neurological disease with a potential to affect functional capacity,
* comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute infections or pneumonia,
* problems which may prevent training such as visual problems and mucositis
* having metastasis to any region (bone etc.)
* having acute hemorrhage in the intracranial and / or lung and other areas
* having any contraindication to exercise training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty-nine allogeneic-HSCT recipients who were at minimum 100 days status post-transplantation, between ages of 18 and 65, under standard medical treatment, transplanted at Bone Marrow Transplantation Unit of University Faculty of Medicine were included. Twenty four severe-fatigued (Fatigue Severity Scale score ≥36) and 25 non-severe-fatigued recipients were compared.Study was approved by local Ethics Committee and informed consent was obtained from all individual participants included in study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Peripheral muscle strength | First day
  Evaluated with a hand-held dynamometer

SECONDARY OUTCOMES:
6-minute walking test | First day
  Evaluated for specifing to functional exercise capacity
Respiratory muscle strength | First day
  Evaluated with a mouth pressure device
Pulmonary function test | First day
  Evaluated with a spirometer
Fatigue Severity Scale | First day
  Fatigue severity was measured using Turkish version of Fatigue Severity Scale. Self-administered questionnaire is consisting of nine questions. An average score is determined on a seven-point scale. Patients mark a number from 1 to 7 for each 9 question which indicates from strong disagreement to strong agreement, respectively. The scale is used in cancer patients.
Modified Medical Research Council Dyspnea scale (MMRC) | First day
  Modified Medical Research Council Dyspnea scale was used to evaluate severity of dyspnea during daily living activities. Dyspnea is graded from zero (absence of dyspnea during strenuous exercise) to four (presence of dyspnea during all daily living activities).
Beck Depression Inventory-II (Turkish version) | First day
  Used for measurement of depression levels
European Organization for Research and Treatment of Cancer QOL Questionnaire (EORTCQOL) | First day
  Quality of life was measured using Turkish version of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 (EORTCQLQ) which is widely used as health related quality of life questionnaire in cancer patients. The cancer-specific questionnaire has 30 questions and incorporates five functional scales, three symptom scales, a global health status and several single items. All item scores are transformed to 0-100. Higher values indicate higher functional/healthy level in functional scales, a higher quality of life level in global health status and increased symptoms in symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD., Study Chair — Gazi University; Meral Boşnak Güçlü, PhD., Study Director — Gazi University; Gülsan Türköz Sucak, PhD., Principal Investigator — Bahçeşehir University
Locations (1):
- Gazi University Faculty of Health Science Department of PhysioTherapy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Result] Paul KL. Rehabilitation and exercise considerations in hematologic malignancies. Am J Phys Med Rehabil. 2011 May;90(5 Suppl 1):S88-94. doi: 10.1097/PHM.0b013e31820be055. PMID 21765268
- [Result] Soutar RL, King DJ. Bone marrow transplantation. BMJ. 1995 Jan 7;310(6971):31-6. doi: 10.1136/bmj.310.6971.31. No abstract available. PMID 7827553
- [Result] Papadopoulos EB, Jakubowski AA. Novel approaches in allogeneic stem cell transplantation. Curr Oncol Rep. 2006 Sep;8(5):325-36. doi: 10.1007/s11912-006-0054-0. PMID 16901394
- [Result] Wulff-Burchfield EM, Jagasia M, Savani BN. Long-term follow-up of informal caregivers after allo-SCT: a systematic review. Bone Marrow Transplant. 2013 Apr;48(4):469-73. doi: 10.1038/bmt.2012.123. Epub 2012 Jun 25. PMID 22732697
- [Result] Polomeni A, Lapusan S, Bompoint C, Rubio MT, Mohty M. The impact of allogeneic-hematopoietic stem cell transplantation on patients' and close relatives' quality of life and relationships. Eur J Oncol Nurs. 2016 Apr;21:248-56. doi: 10.1016/j.ejon.2015.10.011. Epub 2015 Nov 18. PMID 26602410
- [Result] Frodin U, Lotfi K, Fomichov V, Juliusson G, Borjeson S. Frequent and long-term follow-up of health-related quality of life following allogeneic haematopoietic stem cell transplantation. Eur J Cancer Care (Engl). 2015 Nov;24(6):898-910. doi: 10.1111/ecc.12350. Epub 2015 Jul 7. PMID 26156141